CLINICAL TRIAL: NCT00414141
Title: Efficacy and Safety/Tolerability of Grass MATA MPL, a Randomized, Placebo-Controlled, Double-Blind Study
Brief Title: Efficacy and Safety/Tolerability of Grass MATA MPL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Allergy Therapeutics (UK) Ltd., Allergy Therapeutics (UK) Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GrassMATAMPL301
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2009-09

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Allergoid; Specific Immunotherapy
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Grass MATA MPL
  Interventions: Biological: Grass MATA MPL
- 2 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Grass MATA MPL — 4 subcutaneous injections
  Arms: 1
Biological: Placebo — 4 subcutaneous injections
  Other Names: tyrosine solution
  Arms: 2

SUMMARY:
Grass MATA MPL has been developed by Allergy Therapeutics (UK) Ltd. to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to cross reacting grass pollens causing rhinitis and/or conjunctivitis with or without mild to moderate asthma bronchiale. The purpose of this study is to compare the efficacy of Grass MATA MPL versus placebo in grass-allergic subjects following 4 subcutaneous injections of study medication administered before the start of the 2007 grass pollen season.

DETAILED DESCRIPTION:
Grass MATA MPL has been developed by Allergy Therapeutics (UK9 Ltd.to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to cross reacting grass pollens causing rhinitis and/or conjunctivitis with or without mild to moderate asthma bronchiale. Grass MATA MPL is produced as a re-formulation of the Allergy Therapeutics product Pollinex Quattro, which has been used in Europe since 1999 on a 'named patient' basis (with approximately 65,000 treatment courses containing grass pollens).

Grass MATA MPL contains an extract of the 13 grass pollens. This extract is chemically modified with glutaraldehyde to produce the active ingredient, an allergoid. Such modification reduces the reactivity of the extract with IgE antibody. However, a simultaneous reduction in other important immunological properties, such as IgG and T cell reactivity is not seen. The modified extract is adsorbed to L-tyrosine as a depot formulation. MPL®, a purified, detoxified glycolipid derived from the cell walls of Salmonella minnesota, is also included in the current product formulation. This excipient/adjuvant is included to increase the immunogenic effect of the product and to enhance the switch from an allergen-specific TH2 to TH1-like T cell profile.

The current formulation is designed to provide a product that will be efficacious with only 4 injections, in contrast to the longer schedules currently in use with unmodified extracts. The product will also be safer to use than a formulation containing a similar mass of unmodified allergen extract as regards its ability to cause severe local allergic reactions or anaphylaxis, because of its reduced reactivity with IgE antibody. The modification is greater than 75%, so that only a small amount of unmodified allergen is remaining in the product.

The purpose of this study is to compare the efficacy of Grass MATA MPL versus placebo in grass-allergic subjects following 4 subcutaneous injections of study medication administered before the start of the 2007 grass pollen season.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent;
* Are 18 to 59 years of age;
* Have a history of moderate to severe symptoms of seasonal allergic rhinitis and/or conjunctivitis ascribed to grass pollen exposure that required repeated use of antihistamines, nasal steroids, and/or leukotriene modifiers;
* Have a history of moderate to severe symptoms in the past grass pollen season as determined by a score of ≥ 5 on the Disease Severity Questionnaire;
* Have a positive skin prick test to grass pollen mix [wheal (longest diameter) ≥ 5 mm greater than the negative control] and a positive RAST or equivalent test (class ≥ 2) to grass pollen mix;
* Have a positive skin prick test to histamine [wheal (longest diameter) of ≥ 3 mm greater than the negative control];
* Have a negative skin prick test to the negative control (redness with wheal ≤ 2 mm is acceptable);
* Have a forced expiratory volume in 1 second (FEV1) ≥ 80% of predicted, with a FEV1/FVC ratio ≥ 70%;
* Women of childbearing potential must be using a medically acceptable method of birth control [i.e. double barrier method of contraception (e.g., intrauterine device and condom, spermicide and condom), stable hormonal contraceptive for ≥ 90 days prior to the study or if < 90 days additional use of a double barrier method until 90 days reached, sexual abstinence or have a vasectomized partner until study completion], and have a negative β-HCG pregnancy test result at Visits 1 and 2;
* Are able to understand and comply with study instructions;
* Demonstrate proper use of electronic diary with at least 85% compliance (i.e., correct entries for symptoms on 6 of 7 days) during the 1-week period between Visit 1 and Visit 2.

Exclusion Criteria:

* Are pregnant or lactating
* Have asthma requiring the daily use of controller medication;
* Had an emergency room visit or admission for asthma in the 12 months prior to Visit 1;
* Have the presence of secondary alteration at the affected organ (i.e., emphysema, bronchiectasis, nasal polyps, chronic sinusitis);
* Have auto-immune disease (e.g., liver, kidney, thyroid, nervous system);
* Have acute or subacute (historic) atopic dermatitis, chronic dermatitis, urticaria factitia, and/or urticaria due to physical/chemical influence or any other skin conditions which might interfere with the interpretation of the skin prick test results;
* Have a history or presence of diabetes (both insulin dependent and non-dependent), cancer or concomitant illness (e.g., cardiac, metabolic, renal, hepatic, gastrointestinal, dermatologic, venereal, hematologic, neurologic, or psychiatric diseases or disorders) that, in the opinion of the Investigator, would pose a safety risk or compromise the interpretation of efficacy for this grass immunotherapy;
* Have a history of angioedema;
* Have manifest pulmonary or cardiac insufficiency;
* Have current malignant disease;
* Have disorders of tyrosine metabolism (i.e., alcaptonuria, tyrosinemia);
* Have an acute or chronic infection;
* Have any clinically significant abnormal laboratory value (as determined by the Investigator) at Visit 1;
* Perennial Allergens: Have a positive skin prick test [wheal (longest diameter) ≥ 3mm greater than the negative control] at Visit 1 to: house dust mites (Dermatophagoides pteronyssinus and Dermatophagoides farinae), molds (Cladosporium cladosporioides, Alternaria alternata, Penicillium chrysogenum, and Aspergillus fumigatus), or epithelia (cat, dog, and horse). In these cases, a careful history is to be taken and if moderate or severe symptoms are reported when exposed to the aforementioned allergens, the subject is to be excluded. Exception: the source of the allergen (cat, dog, horse) can be avoided for the entire study. Subjects with mild or no symptoms when exposed to the aforementioned allergens during the 3 years prior to Visit 1 will be allowed to enroll. Mild symptoms are defined as: sign/symptom clearly present, but minimal awareness; easily tolerated;
* Only for the USA and Canada:Autumn/Winter Flowering Plant Allergens: Have a positive skin prick test [wheal (longest diameter) ≥ 3mm greater than the negative control] at Visit 1 to: ragweed (Ambrosia sp.) or mountain cedar/mountain juniper (Juniperus ashei). In these cases, a careful history is to be taken and if moderate to severe symptoms are reported when exposed to the aforementioned allergens the subject is to be excluded. Exception: one or both of the listed allergens must not be tested if they are not common to the Investigator's region or, if common to the region, the treatment phase of the study can be initiated at least 30 days after the end of the allergen(s) season. Subjects with mild or no symptoms when exposed to the aforementioned allergens during the 3 years prior to Visit 1 will be allowed to enroll. Mild symptoms are defined as: sign/symptom clearly present, but minimal awareness, easily tolerated;
* Springtime Flowering Plant Allergens: Applies only to subjects living in geographic areas where springtime flowering plant season and grass season overlap and/or when treatment phase cannot be completed at least 30 days prior to the start of the springtime flowering plant season. Otherwise, no testing of the following allergens is necessary; Have a positive skin prick test [wheal (longest diameter) ≥ 3mm greater than the negative control] at Visit 1 to: birch (Betula sp.), oak (Quercus sp.), sycamore/plane (Platanus sp.), beech (Fagus sp.), ash (Fraxinus sp.), or poplar (Populus sp.). In these cases, a careful history is to be taken and if moderate to severe symptoms are reported when exposed to the aforementioned allergens the subject is to be excluded. Subjects with mild or no symptoms when exposed to the aforementioned allergens during the 3 years prior to Visit 1 will be allowed to enroll. Mild symptoms are defined as: sign/symptom clearly present, but minimal awareness, easily tolerated;
* Only for the USA and Canada:Summertime Flowering Plant Allergens: Have a positive skin prick test [wheal (longest diameter) ≥ 3mm greater than the negative control] at Visit 1 to: Bermuda grass (Cynodon dactylon). In these cases, a careful history is to be taken and if moderate to severe symptoms are reported when exposed to the aforementioned allergens the subject is to be excluded. Exception: the listed allergen must not be tested if it is not common to the Investigator's region. Subjects with mild or no symptoms when exposed to the aforementioned allergens during the 3 years prior to Visit 1 will be allowed to enroll. Mild symptoms are defined as: sign/symptom clearly present, but minimal awareness; easily tolerated;
* Have inadequate washout period prior to screening (Visit 1). The following washout periods prior to Visit 1 are acceptable:

  * Oral or parenteral corticosteroids (1 month)
  * Inhaled, ocular or intranasal corticosteroids (1 day)
  * Mast cell stabilizers (7 days)
  * Intranasal or systemic decongestants including cold preparations (1 day)
  * Leukotriene modifiers (7 days)
  * Afrin (oxymetazoline hydrochloride) (14 days)
  * Antihistamines
* Once-daily or twice-daily antihistamines (7 days)
* Short-acting 3 or 4 times a day antihistamines (3 days)
* Hydroxyzine (14 days)

  * H2-blockers (1 day)
  * Other anti-inflammatory, anti-allergy, and any other medications (e.g., anticholinergic agents and tricyclic antidepressants) which, in the opinion of the Investigator, may interfere with the study objectives should be considered on a case-by-case basis
  * Topical skin medications on the forearms (14 days);
* Require use of beta blockers;
* Are unable to receive epinephrine therapy (i.e., use of epinephrine is contraindicated);
* Have a history of anaphylactic reactions to foods, insect venom, exercise, or drugs;
* Have been treated with a preparation containing MPL® within 6 months prior to Visit 1;
* Have diseases with a pathogenesis interfering with the immune response, and who have received medication which could interfere with the results of the study;
* Have a history of allergy, hypersensitivity or intolerance to the excipients of the study medication;
* Have a history of allergy, hypersensitivity or intolerance to study relief medication;
* Have already undergone hyposensitisation therapy with comparable allergen extracts; An exception will be allowed if prior immunotherapy with comparable allergen was successful, symptoms reappeared some time after stopping the immunotherapy, and the immunotherapy was completed ≥ 3 years before Visit 1;
* Have participated in a clinical research trial with a new chemical substance within 4 weeks of Visit 1;
* Are unable or unwilling to cooperate with the Investigator and to comply with the protocol requirements, or not likely to complete the observation periods sufficiently (e.g., 2 weeks holiday abroad during the time of diary recording);
* Have changed residence between geographical regions within the past 3 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1028 (Actual)
Dates: Start 2006-11; Primary Completion 2007-08 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of Grass MATA MPL versus placebo measured by combined allergy symptom + medication scores during 4 peak weeks of grass season | 9 Months

SECONDARY OUTCOMES:
Combined symptom + medication scores, Combined symptoms, Individual symptoms, Relief medication use, Specific immunological changes, quality of life, Health Assessments, Days absent from activities | 9 Months
Adverse events, adverse reactions, clinical labs, ECG, and vitals | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl Jürgen Fischer von Weikersthal-Drachenberg, MD, Study Chair — Allergy Therapeutics
Locations (94):
- United States (65):
  - Asthma & Allergy Associates, PC & Research Center, Colorado Springs, Colorado
  - Colorado Allergy & Asthma Centers, PC, Denver, Colorado
  - Colorado Allergy and Asthma Clinic, PC, Englewood, Colorado
  - Dr. Dreyfus, Waterbury, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Sneeze, Wheeze & Itch Associates, Normal, Illinois
  - The Allergy and Asthma Center, Fort Wayne, Indiana
  - Medical Associates Clinic, Dubuque, Iowa
  - Iowa Clinical Research Corporation, Iowa City, Iowa
  - Kansas City Allergy and Asthma Associates, PA, Overland Park, Kansas
  - Brigham & Women's Hospital, Rheumatology & Immunology, Smith Building Rm 626, Boston, Massachusetts
  - "The Allergy & Arthritis Family Treatment Centers, Gardner, Massachusetts
  - McGovern Allergy Associates, PC, Springfield, Massachusetts
  - Respiratory Medicine Researdh Institute of Michigan, PLC, Ypsilanti, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research Institute, Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Montana Allergy and Asthma 2900 12th Avenue North Suite 302E, Billings, Montana
  - Montana Medical Research, Missoula, Montana
  - Midwest Allegy and Asthma Clinic, Omaha, Nebraska
  - Creighton University - Allergy & Immunology, Omaha, Nebraska
  - Nebraska Medical Research Institute, Papillion, Nebraska
  - Allergy & Asthma Center, Marlboro, New Jersey
  - Princeton Center for Clinical Research Montgomery Professional Center, Skillman, New Jersey
  - The Medical Center at Teaneck, Teaneck, New Jersey
  - Allergy Consultants, PA, Verona, New Jersey
  - Asthma and Allergy Associates, PC, Cortland, New York
  - Asthma and Allergy Associates, PC, Elmira, New York
  - Aair Research Center, Rochester, New York
  - Island Medical Research, PC, Rockville Centre, New York
  - Allergy & Asthma Care Center, Fargo, North Dakota
  - Merit Care Health, Fargo, North Dakota
  - Allergy and Respiratory Center, Canton, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Clinical Research Source, Inc., Perrysburg, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Allergy & Asthma Research Group, Eugene, Oregon
  - Allergy, Asthma and Dermatology Research Center, L.L.C., Lake Oswego, Oregon
  - Clinical Research Institute of Southern, Medford, Oregon
  - Allergy Associates Research Center, LLC, Portland, Oregon
  - MD Office and Research, Altoona, Pennsylvania
  - Asthma & Allergy Research Assoc Presidents House, Chester, Pennsylvania
  - Penn State University Hershey Medical Center, Dept of Medicine, Hershey, Pennsylvania
  - Allergy and Asthma Research of NJ, Philadelphia, Pennsylvania
  - Allergy & Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Allergy Asthma Immunology Clin RI,Ltd, Providence, Rhode Island
  - Asthma Immunology & Allergy, Chattanooga, Tennessee
  - The Allergy, Asthma, and Sinus Center 801 Weisgarber Road, Knoxville, Tennessee
  - Intermountain Clinical Research, Draper, Utah
  - Allergy Associates of Utah, Murray, Utah
  - Clinical Research Specialists of Utah, Spanish Fork, Utah
  - Timber Lane Allergy & Asthma Research, LLC, South Burlington, Vermont
  - Bellingham Asthma And Allergy Associates, Bellingham, Washington
  - Physicians Pharmaceutical Study Services, Everett, Washington
  - Marycliff Allergy Specialists, Spokane, Washington
  - Spokane Allergy & Asthma Clinical Research, Spokane, Washington
  - Pulmonary Consultants, P.L.L.C., Tacoma, Washington
  - Allergy Asthma and Sinus Center, Greenfield, Wisconsin
  - Dean Foundation for Health Research & Education, Inc.Med Reseach Dept., Madison, Wisconsin
  - Advanced Healthcare Clinical Research Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Allergic Diseases, SC, West Allis, Wisconsin
- Austria (4):
  - Universitätsklinik für Umweltdermatologie, Graz
  - Universitätsklinik für Dermatologie und Venerologie, Innsbruck
  - Allgemeines Krankenhaus der Stadt Wien - Universitätsklinik für Dermatologie, Vienna
  - Allergie-Zentrum Wien West, Vienna
- Canada (17):
  - Kelowna Allergy and Respiratory Health Clinic, Kelowna, British Columbia
  - Hamilton Medical Research Group, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario
  - Kanata Allergy Services Ltd., Kanata, Ontario
  - Allied Research International, Mississauga, Ontario
  - Alpha Medical Research Inc., Mississauga, Ontario
  - Niagara Clinical Research, Niagara Falls, Ontario
  - Northgate Medical Clinic, North Bay, Ontario
  - Allergy and Asthma Research Centre, Ottawa, Ontario
  - Filderman R., Toronto, Ontario
  - Knight A., Toronto, Ontario
  - Sussman G., Toronto, Ontario
  - Manna Research, Toronto, Ontario
  - Omnispec Clinical Research, Mirabel, Quebec
  - The McGill University Health Centre, Montreal, Quebec
  - Centre De Recherche Appliquée en Allergie De Québec, Québec, Quebec
  - Q&T Research, Sherbrooke, Quebec
- United Kingdom (8):
  - Birmingham Heartlands Hospital, Birmingham
  - Brighton General Hospital Dept. Respiratory Medicine, Brighton
  - Addenbrookes Hospital, Cambridge
  - Ninewells Hospital and Medical School, Dundee
  - Glenfield Hospital, Leicester
  - Guys Hospital, London
  - Lung Function - Northwest Lung Center, Manchester
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Frew AJ, DuBuske L, Keith PK, Corrigan CJ, Aberer W, Fischer von Weikersthal-Drachenberg KJ. Assessment of specific immunotherapy efficacy using a novel placebo score-based method. Ann Allergy Asthma Immunol. 2012 Nov;109(5):342-347.e1. doi: 10.1016/j.anai.2012.08.013. PMID 23062390